CLINICAL TRIAL: NCT01358110
Title: Emergency Department-Based Palliative Care for Advanced Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: GCO 08-1234
Record Dates: First submitted 2011-05-19; First posted 2011-05-23 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Advanced Cancer; Metastatic Cancer
Keywords: palliative care; cancer; emergency medicine; end- of- life care
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early palliative care consultation (Experimental): Early palliative care consultation for ED patients with advanced cancer.
  Interventions: Other: Early palliative care consultation
- Care as usual (Other): Care as usual, may or may not receive palliative care consultation
  Interventions: Other: Care as usual

INTERVENTIONS:
Other: Early palliative care consultation — Patients will have symptoms assessed, have goals of care discussion with family and team present, and surrogate designated, as well as coordination of care and home services.
  Arms: Early palliative care consultation
Other: Care as usual — Standard care as usual which may or may not include palliative care consultation
  Arms: Care as usual

SUMMARY:
The purpose of this study is to: 1) identify the palliative care needs of Emergency Department patients with advanced cancer, and determine if these needs can be rapidly assessed in the ED; 2) determine whether early palliative care consultation improves survival, quality of life and other burdensome symptoms and decreases utilization as compared to usual care.

DETAILED DESCRIPTION:
As the population ages, the number of individual living with cancer will continue to rise, and the number of Emergency Department (ED) visits for this population will continue to increase. Cancer patients visit EDs because symptoms, such as pain or vomiting, can't be controlled at home, in an assisted living facility, or in their provider's office. The ED is often the only place that can provide the necessary treatments as well as immediate access to technologically advanced testing for those with cancer. However, palliative care (PC) services, such as relief of burdensome symptoms), attention to spiritual or social concerns, and establishing goals of care, is not standard care in the ED outside of a few medical centers. Most patients do not have well-defined goals of care, and are often subjected to painful and marginally effective tests and procedures, not because they are consistent with their goals but because it is less time-consuming than discussing other options and has less perceived legal risk. Until recently little emphasis has been placed on education, research, or guidelines for the delivery of PC services in this important setting. While emergency providers could provide some of these services themselves, knowledge and skills regarding PC as well as staffing are currently inadequate to provide comprehensive services. In addition to further decreasing days spent in the hospital and health care costs, consultation by a PC team for ED cancer patients might also reduce pain and other symptoms, aid in complex medical decision-making regarding testing and treatments, and facilitate transfer to hospice or home with visiting nurse services. To enable PC consultation for ED cancer patients, the investigators will first determine who could benefit from emergent consultation, what services they need, and what characteristics of emergency providers and hospitals are preventing them from being offered. To determine what affect PC consultation for patients with advanced cancer has on symptoms, discussions with patients and families about goals of care, and how long patients spend in the ED, the investigators will then randomly assign 200 ED cancer patients to targeted PC consultation versus usual or standard care.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years age
* Speak English or Spanish
* ED patient with an advanced solid malignancy

Exclusion Criteria:

* Have already been seen by palliative care team
* Cognitive deficits
* Children or adolescents
* No confirmed history of active cancer
* Do not speak English or Spanish
* Reside outside the US

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2011-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Quality of life and quality of mental health at 6 weeks and 12 weeks as compared from baseline | at baseline, 6 weeks and 12 weeks
  Comparison of life and quality of mental health from baseline to 6 weeks and 12 weeks.

SECONDARY OUTCOMES:
Inpatient costs per day/cost of stay during hospitalization | 6 months after hospital discharge
  Costs per day during incident admission and total cost of entire incident hospital stay
Hospital length of stay | 6 months after hospital discharge
  Number of days hospitalized for incident admission: i.e., date of admission and date of discharge, difference between those two dates.
Survival | at time of enrollment
  Survival days from day of enrollment to day of death or study termination
Readmissions within 6 months of discharge | 6 months from hospital discharge
Repeat visits to the ED in 6 months | 6 months from hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Corita Grudzen, MD, MSHS, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Wiencke JK, Zheng S, Lafuente A, Lafuente MJ, Grudzen C, Wrensch MR, Miike R, Ballesta A, Trias M. Aberrant methylation of p16INK4a in anatomic and gender-specific subtypes of sporadic colorectal cancer. Cancer Epidemiol Biomarkers Prev. 1999 Jun;8(6):501-6. PMID 10385139
- [Background] Grudzen CR, Liddicoat R, Hoffman JR, Koenig W, Lorenz KA, Asch SM. Developing quality indicators for the appropriateness of resuscitation in prehospital atraumatic cardiac arrest. Prehosp Emerg Care. 2007 Oct-Dec;11(4):434-42. doi: 10.1080/10903120701536925. PMID 17907029
- [Background] Chan GK. End-of-life models and emergency department care. Acad Emerg Med. 2004 Jan;11(1):79-86. doi: 10.1197/j.aem.2003.07.019. PMID 14709435
- [Background] McCusker J, Karp I, Cardin S, Durand P, Morin J. Determinants of emergency department visits by older adults: a systematic review. Acad Emerg Med. 2003 Dec;10(12):1362-70. doi: 10.1111/j.1553-2712.2003.tb00011.x. PMID 14644789
- [Background] Burge F, Lawson B, Johnston G. Family physician continuity of care and emergency department use in end-of-life cancer care. Med Care. 2003 Aug;41(8):992-1001. doi: 10.1097/00005650-200308000-00012. PMID 12886178
- [Background] A controlled trial to improve care for seriously ill hospitalized patients. The study to understand prognoses and preferences for outcomes and risks of treatments (SUPPORT). The SUPPORT Principal Investigators. JAMA. 1995 Nov 22-29;274(20):1591-8. PMID 7474243
- [Background] Mohanty SA SS, Bodukum VK,Grudzen CR, Lorenz K, Asch SM. Assessing the Need for Integration of Palliative Care in a Public Sector Emergency Department. Paper presented at: Academy Health2008; Washington D.C.
- [Background] Mahony SO, Blank A, Simpson J, Persaud J, Huvane B, McAllen S, Davitt M, McHugh M, Hutcheson A, Karakas S, Higgins P, Selwyn P. Preliminary report of a palliative care and case management project in an emergency department for chronically ill elderly patients. J Urban Health. 2008 May;85(3):443-51. doi: 10.1007/s11524-008-9257-z. PMID 18363108
- [Background] Alpert HR, Emanuel L. Comparing utilization of life-sustaining treatments with patient and public preferences. J Gen Intern Med. 1998 Mar;13(3):175-81. doi: 10.1046/j.1525-1497.1998.00052.x. PMID 9541374
- [Background] Marco CA, Bessman ES, Schoenfeld CN, Kelen GD. Ethical issues of cardiopulmonary resuscitation: current practice among emergency physicians. Acad Emerg Med. 1997 Sep;4(9):898-904. doi: 10.1111/j.1553-2712.1997.tb03816.x. PMID 9305432
- [Background] Lunney JR, Lynn J, Foley DJ, Lipson S, Guralnik JM. Patterns of functional decline at the end of life. JAMA. 2003 May 14;289(18):2387-92. doi: 10.1001/jama.289.18.2387. PMID 12746362
- [Background] Covinsky KE, Eng C, Lui LY, Sands LP, Yaffe K. The last 2 years of life: functional trajectories of frail older people. J Am Geriatr Soc. 2003 Apr;51(4):492-8. doi: 10.1046/j.1532-5415.2003.51157.x. PMID 12657068
- [Background] Partnership for Solutions. Chronic Conditions: Making the Case for Ongoing Care. Baltimore: Johns Hopkins University;2002.
- [Background] Greenlee RT, Hill-Harmon MB, Murray T, Thun M. Cancer statistics, 2001. CA Cancer J Clin. 2001 Jan-Feb;51(1):15-36. doi: 10.3322/canjclin.51.1.15. PMID 11577478
- [Background] McKinley ED, Garrett JM, Evans AT, Danis M. Differences in end-of-life decision making among black and white ambulatory cancer patients. J Gen Intern Med. 1996 Nov;11(11):651-6. doi: 10.1007/BF02600155. PMID 9120650
- [Background] Field MJ, Cassel CK. Approaching death: improving care at the end of life. Health Prog. 2011 Jan-Feb;92(1):25. No abstract available. PMID 21306019
- [Background] Institute of Medicine (US) and National Research Council (US) National Cancer Policy Board; Foley KM, Gelband H, editors. Improving Palliative Care for Cancer. Washington (DC): National Academies Press (US); 2001. Available from http://www.ncbi.nlm.nih.gov/books/NBK223535/ PMID 25057564
- [Background] Institute of Medicine (U.S.). Committee on Palliative and End-of-Life Care for Children and Their Families. Ethical and legal issues. Washington, D.C.: Institute of Medicine, National Academies Press; 2003.
- [Background] NIH State-of-the-Science Conference Statement on improving end-of-life care. NIH Consens State Sci Statements. 2004 Dec 6-8;21(3):1-26. PMID 17308546
- [Background] Lubitz JD, Riley GF. Trends in Medicare payments in the last year of life. N Engl J Med. 1993 Apr 15;328(15):1092-6. doi: 10.1056/NEJM199304153281506. PMID 8455667
- [Background] American Cancer Society. Cancer Facts and Figures. 2008; http://www.cancer.org/docroot/STT/content/STT_1x_Cancer_Facts_and_Figures_2008.asp. Accessed October 2, 2008.
- [Background] DeFrances CJ, Hall MJ. 2002 National Hospital Discharge Survey. Adv Data. 2004 May 21;(342):1-29. PMID 15174387
- [Background] American Academy of Hospice and Palliative Medicine; Center to Advance Palliative Care; Hospice and Palliative Nurses Association; Last Acts Partnership; National Hospice and Palliative Care Organization. National Consensus Project for Quality Palliative Care: Clinical Practice Guidelines for quality palliative care, executive summary. J Palliat Med. 2004 Oct;7(5):611-27. doi: 10.1089/jpm.2004.7.611. No abstract available. PMID 15588352
- [Background] Block SD. Perspectives on care at the close of life. Psychological considerations, growth, and transcendence at the end of life: the art of the possible. JAMA. 2001 Jun 13;285(22):2898-905. doi: 10.1001/jama.285.22.2898. PMID 11401612
- [Background] Portenoy RK, Frager G. Pain management: pharmacological approaches. Cancer Treat Res. 1999;100:1-29. doi: 10.1007/978-1-4615-5003-7_1. No abstract available. PMID 10645494
- [Background] Bruera E. ABC of palliative care. Anorexia, cachexia, and nutrition. BMJ. 1997 Nov 8;315(7117):1219-22. doi: 10.1136/bmj.315.7117.1219. No abstract available. PMID 9393230
- [Background] Tulsky JA. Doctor-Patient Communication. In: Morrison RS, Meier DE, eds. Geriatric Palliative Care. New York: Oxford University Press; 2003.
- [Background] Fallowfield L, Jenkins V. Communicating sad, bad, and difficult news in medicine. Lancet. 2004 Jan 24;363(9405):312-9. doi: 10.1016/S0140-6736(03)15392-5. PMID 14751707
- [Background] Emanuel EJ, Fairclough DL, Slutsman J, Emanuel LL. Understanding economic and other burdens of terminal illness: the experience of patients and their caregivers. Ann Intern Med. 2000 Mar 21;132(6):451-9. doi: 10.7326/0003-4819-132-6-200003210-00005. PMID 10733444
- [Background] Tolle SW, Tilden VP, Rosenfeld AG, Hickman SE. Family reports of barriers to optimal care of the dying. Nurs Res. 2000 Nov-Dec;49(6):310-7. doi: 10.1097/00006199-200011000-00003. PMID 11093695
- [Background] Quill TE. Perspectives on care at the close of life. Initiating end-of-life discussions with seriously ill patients: addressing the "elephant in the room". JAMA. 2000 Nov 15;284(19):2502-7. doi: 10.1001/jama.284.19.2502. PMID 11074781
- [Background] Lo B, Quill T, Tulsky J. Discussing palliative care with patients. ACP-ASIM End-of-Life Care Consensus Panel. American College of Physicians-American Society of Internal Medicine. Ann Intern Med. 1999 May 4;130(9):744-9. No abstract available. PMID 10357694
- [Background] Quill TE, Arnold RM, Platt F. "I wish things were different": expressing wishes in response to loss, futility, and unrealistic hopes. Ann Intern Med. 2001 Oct 2;135(7):551-5. doi: 10.7326/0003-4819-135-7-200110020-00022. No abstract available. PMID 11578166
- [Background] von Gunten CF, Ferris FD, Emanuel LL. The patient-physician relationship. Ensuring competency in end-of-life care: communication and relational skills. JAMA. 2000 Dec 20;284(23):3051-7. doi: 10.1001/jama.284.23.3051. PMID 11122596
- [Background] Singer PA, Martin DK, Kelner M. Quality end-of-life care: patients' perspectives. JAMA. 1999 Jan 13;281(2):163-8. doi: 10.1001/jama.281.2.163. PMID 9917120
- [Background] Bass DM, Noelker LS, Rechlin LR. The moderating influence of service use on negative caregiving consequences. J Gerontol B Psychol Sci Soc Sci. 1996 May;51(3):S121-31. doi: 10.1093/geronb/51b.3.s121. PMID 8620359
- [Background] Levine C. The loneliness of the long-term care giver. N Engl J Med. 1999 May 20;340(20):1587-90. doi: 10.1056/NEJM199905203402013. No abstract available. PMID 10332025
- [Background] McClain CS, Rosenfeld B, Breitbart W. Effect of spiritual well-being on end-of-life despair in terminally-ill cancer patients. Lancet. 2003 May 10;361(9369):1603-7. doi: 10.1016/S0140-6736(03)13310-7. PMID 12747880
- [Background] Meier DE, Thar W, Jordan A, Goldhirsch SL, Siu A, Morrison RS. Integrating case management and palliative care. J Palliat Med. 2004 Feb;7(1):119-34. doi: 10.1089/109662104322737395. PMID 15000796
- [Background] Bass DM, Bowman K, Noelker LS. The influence of caregiving and bereavement support on adjusting to an older relative's death. Gerontologist. 1991 Feb;31(1):32-42. doi: 10.1093/geront/31.1.32. PMID 2007473
- [Background] Billings JA. What is palliative care? J Palliat Med. 1998 Spring;1(1):73-81. doi: 10.1089/jpm.1998.1.73. No abstract available. PMID 15859874
- [Background] Meier DE, Morrison RS, Cassel CK. Improving palliative care. Ann Intern Med. 1997 Aug 1;127(3):225-30. doi: 10.7326/0003-4819-127-3-199708010-00008. PMID 9245229
- [Background] Morrison RS, Meier DE. Clinical practice. Palliative care. N Engl J Med. 2004 Jun 17;350(25):2582-90. doi: 10.1056/NEJMcp035232. No abstract available. PMID 15201415
- [Background] National Quality Forum. A national framework and preferred practices for palliative and hospice care quality : a consensus report. Washington, DC: National Quality Forum; 2006.
- [Background] Clinical Practice Guidelines for Quality Palliative Care. National Consensus Project for Quality Palliative Care 2004; www.nationalconsensusproject.org. Accessed November 8, 2009.
- [Background] Byock I. Completing the continuum of cancer care: integrating life-prolongation and palliation. CA Cancer J Clin. 2000 Mar-Apr;50(2):123-32. doi: 10.3322/canjclin.50.2.123. PMID 10870488
- [Background] Center for the Evaluative Clinical Sciences. Dartmouth Atlas of Health Care. 1999; 2001:http://www.dartmouthatlas.org/atlases/2006_Atlas_Exec_Summary.pdf.
- [Background] Lynn J, Wilkinson AM. Quality end of life care: the case for a MediCaring demonstration. Hosp J. 1998;13(1-2):151-63. doi: 10.1080/0742-969x.1998.11882895. PMID 9644400
- [Background] Lynn J. Perspectives on care at the close of life. Serving patients who may die soon and their families: the role of hospice and other services. JAMA. 2001 Feb 21;285(7):925-32. doi: 10.1001/jama.285.7.925. PMID 11180736
- [Background] Lynn J. Learning to care for people with chronic illness facing the end of life. JAMA. 2000 Nov 15;284(19):2508-11. doi: 10.1001/jama.284.19.2508. No abstract available. PMID 11074783
- [Background] Eng C, Pedulla J, Eleazer GP, McCann R, Fox N. Program of All-inclusive Care for the Elderly (PACE): an innovative model of integrated geriatric care and financing. J Am Geriatr Soc. 1997 Feb;45(2):223-32. doi: 10.1111/j.1532-5415.1997.tb04513.x. PMID 9033525
- [Background] Center to Advance Palliative Care. A Guide to Developing a Hospital-Based Palliative Care Program. New York: Center to Advance Palliative Care; 2004.
- [Background] von Gunten CF. Secondary and tertiary palliative care in US hospitals. JAMA. 2002 Feb 20;287(7):875-81. doi: 10.1001/jama.287.7.875. PMID 11851580
- [Background] McMillan SC, Small BJ. Using the COPE intervention for family caregivers to improve symptoms of hospice homecare patients: a clinical trial. Oncol Nurs Forum. 2007 Mar;34(2):313-21. doi: 10.1188/07.ONF.313-321. PMID 17573295
- [Background] Brumley R, Enguidanos S, Jamison P, Seitz R, Morgenstern N, Saito S, McIlwane J, Hillary K, Gonzalez J. Increased satisfaction with care and lower costs: results of a randomized trial of in-home palliative care. J Am Geriatr Soc. 2007 Jul;55(7):993-1000. doi: 10.1111/j.1532-5415.2007.01234.x. PMID 17608870
- [Background] Rummans TA, Clark MM, Sloan JA, Frost MH, Bostwick JM, Atherton PJ, Johnson ME, Gamble G, Richardson J, Brown P, Martensen J, Miller J, Piderman K, Huschka M, Girardi J, Hanson J. Impacting quality of life for patients with advanced cancer with a structured multidisciplinary intervention: a randomized controlled trial. J Clin Oncol. 2006 Feb 1;24(4):635-42. doi: 10.1200/JCO.2006.06.209. PMID 16446335
- [Background] Engelhardt JB, McClive-Reed KP, Toseland RW, Smith TL, Larson DG, Tobin DR. Effects of a program for coordinated care of advanced illness on patients, surrogates, and healthcare costs: a randomized trial. Am J Manag Care. 2006 Feb;12(2):93-100. PMID 16464138
- [Background] Casarett D, Karlawish J, Morales K, Crowley R, Mirsch T, Asch DA. Improving the use of hospice services in nursing homes: a randomized controlled trial. JAMA. 2005 Jul 13;294(2):211-7. doi: 10.1001/jama.294.2.211. PMID 16014595
- [Background] Hughes SL, Weaver FM, Giobbie-Hurder A, Manheim L, Henderson W, Kubal JD, Ulasevich A, Cummings J; Department of Veterans Affairs Cooperative Study Group on Home-Based Primary Care. Effectiveness of team-managed home-based primary care: a randomized multicenter trial. JAMA. 2000 Dec 13;284(22):2877-85. doi: 10.1001/jama.284.22.2877. PMID 11147984
- [Background] Moore S, Corner J, Haviland J, Wells M, Salmon E, Normand C, Brada M, O'Brien M, Smith I. Nurse led follow up and conventional medical follow up in management of patients with lung cancer: randomised trial. BMJ. 2002 Nov 16;325(7373):1145. doi: 10.1136/bmj.325.7373.1145. PMID 12433764
- [Background] Ciemins EL, Blum L, Nunley M, Lasher A, Newman JM. The economic and clinical impact of an inpatient palliative care consultation service: a multifaceted approach. J Palliat Med. 2007 Dec;10(6):1347-55. doi: 10.1089/jpm.2007.0065. PMID 18095814
- [Background] Cowan JD. Hospital charges for a community inpatient palliative care program. Am J Hosp Palliat Care. 2004 May-Jun;21(3):177-90. doi: 10.1177/104990910402100306. PMID 15188917
- [Background] Norton SA, Hogan LA, Holloway RG, Temkin-Greener H, Buckley MJ, Quill TE. Proactive palliative care in the medical intensive care unit: effects on length of stay for selected high-risk patients. Crit Care Med. 2007 Jun;35(6):1530-5. doi: 10.1097/01.CCM.0000266533.06543.0C. PMID 17452930
- [Background] Twaddle ML, Maxwell TL, Cassel JB, Liao S, Coyne PJ, Usher BM, Amin A, Cuny J. Palliative care benchmarks from academic medical centers. J Palliat Med. 2007 Feb;10(1):86-98. doi: 10.1089/jpm.2006.0048. PMID 17298257
- [Background] O'Mahony S, Blank AE, Zallman L, Selwyn PA. The benefits of a hospital-based inpatient palliative care consultation service: preliminary outcome data. J Palliat Med. 2005 Oct;8(5):1033-9. doi: 10.1089/jpm.2005.8.1033. PMID 16238516
- [Background] Hanson LC, Usher B, Spragens L, Bernard S. Clinical and economic impact of palliative care consultation. J Pain Symptom Manage. 2008 Apr;35(4):340-6. doi: 10.1016/j.jpainsymman.2007.06.008. Epub 2008 Feb 8. PMID 18261877
- [Background] Penrod JD, Deb P, Luhrs C, Dellenbaugh C, Zhu CW, Hochman T, Maciejewski ML, Granieri E, Morrison RS. Cost and utilization outcomes of patients receiving hospital-based palliative care consultation. J Palliat Med. 2006 Aug;9(4):855-60. doi: 10.1089/jpm.2006.9.855. PMID 16910799
- [Background] Axelsson B, Christensen SB. Evaluation of a hospital-based palliative support service with particular regard to financial outcome measures. Palliat Med. 1998 Jan;12(1):41-9. doi: 10.1191/026921698671336362. PMID 9616458
- [Background] Hughes SL, Cummings J, Weaver F, Manheim L, Braun B, Conrad K. A randomized trial of the cost effectiveness of VA hospital-based home care for the terminally ill. Health Serv Res. 1992 Feb;26(6):801-17. PMID 1737710
- [Background] Zimmer JG, Groth-Juncker A, McCusker J. Effects of a physician-led home care team on terminal care. J Am Geriatr Soc. 1984 Apr;32(4):288-92. doi: 10.1111/j.1532-5415.1984.tb02023.x. PMID 6707409
- [Background] Kane RL, Wales J, Bernstein L, Leibowitz A, Kaplan S. A randomised controlled trial of hospice care. Lancet. 1984 Apr 21;1(8382):890-4. doi: 10.1016/s0140-6736(84)91349-7. PMID 6143195
- [Background] Jordhoy MS, Fayers P, Loge JH, Ahlner-Elmqvist M, Kaasa S. Quality of life in palliative cancer care: results from a cluster randomized trial. J Clin Oncol. 2001 Sep 15;19(18):3884-94. doi: 10.1200/JCO.2001.19.18.3884. PMID 11559726
- [Background] McCorkle R, Benoliel JQ, Donaldson G, Georgiadou F, Moinpour C, Goodell B. A randomized clinical trial of home nursing care for lung cancer patients. Cancer. 1989 Sep 15;64(6):1375-82. doi: 10.1002/1097-0142(19890915)64:63.0.co;2-6. PMID 2670188
- [Background] Rabow MW, Dibble SL, Pantilat SZ, McPhee SJ. The comprehensive care team: a controlled trial of outpatient palliative medicine consultation. Arch Intern Med. 2004 Jan 12;164(1):83-91. doi: 10.1001/archinte.164.1.83. PMID 14718327
- [Background] Pantilat SZ, Billings JA. Prevalence and structure of palliative care services in California hospitals. Arch Intern Med. 2003 May 12;163(9):1084-8. doi: 10.1001/archinte.163.9.1084. PMID 12742807
- [Background] Billings JA, Pantilat S. Survey of palliative care programs in United States teaching hospitals. J Palliat Med. 2001 Fall;4(3):309-14. doi: 10.1089/109662101753123913. PMID 11596541
- [Background] Pan CX, Morrison RS, Meier DE, Natale DK, Goldhirsch SL, Kralovec P, Cassel CK. How prevalent are hospital-based palliative care programs? Status report and future directions. J Palliat Med. 2001 Fall;4(3):315-24. doi: 10.1089/109662101753123922. PMID 11596542
- [Background] Morrison RS, Maroney-Galin C, Kralovec PD, Meier DE. The growth of palliative care programs in United States hospitals. J Palliat Med. 2005 Dec;8(6):1127-34. doi: 10.1089/jpm.2005.8.1127. PMID 16351525
- [Background] Morrison RS, Penrod JD, Cassel JB, Caust-Ellenbogen M, Litke A, Spragens L, Meier DE; Palliative Care Leadership Centers' Outcomes Group. Cost savings associated with US hospital palliative care consultation programs. Arch Intern Med. 2008 Sep 8;168(16):1783-90. doi: 10.1001/archinte.168.16.1783. PMID 18779466
- [Background] Osta BE, Palmer JL, Paraskevopoulos T, Pei BL, Roberts LE, Poulter VA, Chacko R, Bruera E. Interval between first palliative care consult and death in patients diagnosed with advanced cancer at a comprehensive cancer center. J Palliat Med. 2008 Jan-Feb;11(1):51-7. doi: 10.1089/jpm.2007.0103. PMID 18370893
- [Background] Scalise D. The American Hospital Association 2004 NOVA Award winners. Trustee. 2004 Sep;57(8):21-5. No abstract available. PMID 15597503
- [Background] Goldsmith B, Dietrich J, Du Q, Morrison RS. Variability in access to hospital palliative care in the United States. J Palliat Med. 2008 Oct;11(8):1094-102. doi: 10.1089/jpm.2008.0053. PMID 18831653
- [Background] Improving Palliative Care for Cancer. Washington D.C.: Institute of Medicine and National Research Council; National Academy Press; 2001.
- [Background] American Cancer Society: Strategic Plan and Progress Report. 2007; http://www.cancer.org/downloads/AA/2007_Strategic_Plan_Progress_Report.pdf. Accessed October 6, 2008.
- [Background] Donnelly S, Walsh D. The symptoms of advanced cancer. Semin Oncol. 1995 Apr;22(2 Suppl 3):67-72. PMID 7537907
- [Derived] Grudzen CR, Richardson LD, Johnson PN, Hu M, Wang B, Ortiz JM, Kistler EA, Chen A, Morrison RS. Emergency Department-Initiated Palliative Care in Advanced Cancer: A Randomized Clinical Trial. JAMA Oncol. 2016 May 1;2(5):591-598. doi: 10.1001/jamaoncol.2015.5252. PMID 26768772
- [Derived] Kistler EA, Sean Morrison R, Richardson LD, Ortiz JM, Grudzen CR. Emergency department-triggered palliative care in advanced cancer: proof of concept. Acad Emerg Med. 2015 Feb;22(2):237-9. doi: 10.1111/acem.12573. Epub 2015 Jan 29. PMID 25639187
- [Derived] Kandarian B, Morrison RS, Richardson LD, Ortiz J, Grudzen CR. Emergency department-initiated palliative care for advanced cancer patients: protocol for a pilot randomized controlled trial. Trials. 2014 Jun 25;15:251. doi: 10.1186/1745-6215-15-251. PMID 24962353